CLINICAL TRIAL: NCT00169962
Title: Use of Aerosolized rhDNase (Pulmozyme®) in Emergency Department Adults With Refractory Acute Asthma: A Pilot Study
Brief Title: Study of Pulmozyme to Treat Severe Asthma Episodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert A Silverman, Physician, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03.05.086
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: acute disease
MeSH Terms: conditions — Asthma; Acute Disease | interventions — dornase alfa

INTERVENTIONS:
Drug: rhDNAse (pulmozyme)

SUMMARY:
Even with current standard ED treatments 20-25% of patients presenting to the ED with an acute asthma episode will still require hospitalization. For patients unresponsive to beta-agonists the admit rates will be higher. Of those well enough to be discharged from the ED nearly 30% will relapse within one month. More than 5,000 patients with asthma still die each year in the USA. For patients who do not respond to beta-agonists, there are relatively few treatment options for rapid improvement of symptoms and pulmonary function. Presumably, mucous secretion and plugging play an important role in the pathogenesis of severe asthma unresponsive to beta-agonists. The use of agents to promote clearance of intra-luminal secretions and mucous plugs may represent an important advance in the management of acutely ill asthmatics, both to hasten recovery and prevent deterioration in the acute care setting and to prevent relapse after discharge from the ED.

OBJECTIVES

2.1 Study Hypothesis: rhDNAse can be safely used in patients presenting to the Emergency Department with acute moderate-severe asthma who do not have adequate responses to beta-agonists

Project Specific Aim: This is a pilot study to determine the safety of three different doses of pulmozyme® (2.5mg, 5.0mg and 7.5mg) in patients presenting to the ED with acute asthma. In addition to safety trends for improvement in pulmonary function and clinical outcomes will be monitored and data analyzed. Based on the safety profile and observable responses to treatment, this information may be used to develop larger trials to determine the efficacy and dosing strategy for treating acutely ill asthmatics with rhDNAse.

ELIGIBILITY:
Inclusion Criteria:

acute asthma FEV1<60% post-standard care age 18-55 years -

Exclusion Criteria:

other chronic lung illness pregnancy -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
FEV1

SECONDARY OUTCOMES:
Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Silverman, MD, Principal Investigator — LIJMC
Locations (1):
- LIJMC, Queens, New York, United States

REFERENCES:
- [Derived] Silverman RA, Foley F, Dalipi R, Kline M, Lesser M. The use of rhDNAse in severely ill, non-intubated adult asthmatics refractory to bronchodilators: a pilot study. Respir Med. 2012 Aug;106(8):1096-102. doi: 10.1016/j.rmed.2012.04.002. Epub 2012 May 12. PMID 22580235